CLINICAL TRIAL: NCT05107804
Title: Effects of Moderate Aerobic Exercise Combined With Caloric Restriction on Circulating Estrogens and IGF-I in Premenopausal Women
Brief Title: Energy Restriction and Hormones in Premenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); United States Department of Defense (U.S. Federal Agency); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Nancy Williams, Professor and Head, Department of Kinesiology, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01M0088; M01RR010732 (NIH); DAMD 17-01-1-0361 (Other Grant/Funding Number: Department of Defense); DAMD 17-01-109360 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2021-10-06; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Menstruation Disturbances; Luteal Phase Defect
Keywords: Energy Balance; Menstrual Cycle Disturbance; Luteal Phase Defect; Menstruation Disturbances; Pathologic Processes
MeSH Terms: conditions — Menstruation Disturbances; Pathologic Processes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise with caloric-restriction (Experimental): Exercise: Participants engaged in supervised exercise training sessions (to expend ~20% of baseline energy needs) in Noll Laboratory; 4 times per week.
  Diet: Participants consumed meals in the General Clinical Research Center metabolic kitchen that reduced dietary intake 20-35% of baseline energy needs. Diet composition was 55% carbohydrates, 30% fat, and 15% protein.
  Interventions: Other: Exercise+CR
- Light Conditioning (reference group) (Active Comparator): Exercise: Participants engaged in supervised exercise training sessions (to expend ~10% of baseline energy needs) in Noll Laboratory; 1-2 times per week.
  Diet: Participants consumed meals in the General Clinical Research Center metabolic kitchen that had calories sufficient to maintain body weight and additional calories to remain in energy balance. Diet composition was 55% carbohydrates, 30% fat, and 15% protein.
  Interventions: Other: Light Conditioning

INTERVENTIONS:
Other: Exercise+CR — Exercise with caloric-restriction
  Arms: Exercise with caloric-restriction
Other: Light Conditioning — Light Conditioning Exercise
  Arms: Light Conditioning (reference group)

SUMMARY:
A growing body of epidemiological and biological evidence strongly suggests that physical activity may reduce the risk of breast cancer. Although the mechanism remains unclear, possible links between reduced risk and exercise include favorable alterations in body composition and positive changes in the hormonal milieu. One hormonal biomarker of breast cancer, circulating estrogen, is postulated to be reduced by chronic physical activity, presumably due to disruptive effects of exercise upon menstrual cyclicity, and the potential for loss of body fat with subsequent reductions in the peripheral biosynthesis of circulating estrogens. Although studies have shown that chronic exercise can reduce circulating estrogen, we know little about the magnitude and duration of exposure to an energy deficit required for these changes. Additionally, no studies have addressed the degree to which peripheral production of estrone, versus the ovarian production of estradiol, is altered with exercise that promotes weight/fat loss. A second biomarker of breast cancer, insulin-like growth factor-1 (IGF-1), is presumably increased with exercise but reduced with exercise if energy balance is negative. No prospective studies have addressed whether a moderate aerobic exercise program that results in weight loss will lead to significant changes in IGF-I levels, particularly in individuals of differing initial energy stores.

Metabolic energy availability is an important contributing factor in the development of reproductive cancers. However, current methods for assessing energy availability, which include anthropometric measures, calculations of energy balance, evaluation of various serum and urinary biomarkers are prone to measurement error, not sensitive to alterations in energy availability, and are sometimes affected by disease states. The current project includes the introduction of a novel approach to estimating energy status by measuring metabolic hormones in plasma: insulin, IGF-I, insulin-like growth factor binding protein-3 (IGFBP-3) and leptin.

This study tested whether a program of moderate aerobic exercise that is combined with a moderate level of dietary restriction would result in significant decreases in two biomarkers of breast cancer, circulating estrogens and IGF-I.

DETAILED DESCRIPTION:
This study used a randomized prospective design (block; 3:1 allocation) to test the effects of a four month (four menstrual cycles) intervention of moderate aerobic exercise (4 times per week, 60 minutes/session) combined with caloric restriction designed to produce a weekly energy deficit of -20%. The aims of the study were: 1) To test the hypothesis that a moderate level of low energy availability created through a combination of exercise and caloric restriction will lower circulating estrogens and IGF-I; 2) To test the hypothesis that exercise-induced decreases in body fat will contribute substantially to the lowering of circulating estrogens changes with training; 3) To validate a novel method of assessing energy status that represents an improvement of existing.

Eumenorrheic, untrained women between 25-40 years (n=47) were randomly assigned to one of two treatments groups: exercise with caloric-restriction (EX+CR; n=36) or light conditioning reference (LC; n=11) groups. To determine treatment effects on circulating estrogens, reproductive function and IGF-I, both serum and urinary levels of hormones were monitored for a control period of 2 months (2 menstrual cycles), i.e., Screening and Baseline, followed the 4 month (4 menstrual cycles: intervention 1-4) experimental period. The exercise/diet intervention began on the first day of the third month (menstrual cycle) and continue for four menstrual cycles thereafter (intervention 1, 2, 3, and 4). A post-study measurement was taken during cycles days 1-7 of the seventh menstrual cycle.

Baseline energy needs were assessed during the baseline cycle. Resting metabolic rate and non-exercise physical activity were added to determine a caloric need for the day. Caloric intake was supervised throughout the entire study, and meals were comprised of 55% carbohydrates, 30% fat, and 15% protein. Exercise training was supervised, and maximal aerobic capacity (VO2max) was calculated. Menstrual status was assessed through analysis of daily urinary metabolites of estrone-1-glucuronide (E1G), pregnanediol glucuronide (PdG), and midcycle luteinizing hormone (LH). Underwater weighing and a digital scale were used to assess body composition, and fasting blood samples were collected to assess metabolic hormones.

ELIGIBILITY:
Inclusion Criteria:

* Weight 50-90 kg
* BMI 18-35 kg/m2
* Nonsmoking
* <1 hour/week of purposeful aerobic exercise for the past 6 months
* Gynecological age ≥10 years
* Documentation of at least two ovulatory menstrual cycles during screening.

Exclusion Criteria:

* History of serious medical conditions
* Medication use that would alter metabolic hormone levels
* Significant weight loss/gain (±2.3 kg) in the last year
* Current evidence of disordered eating or history of an eating disorder
* Taking exogenous hormonal contraceptives for the past 6 month
* Smoking

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2001-03 (Actual); Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Change in estrogen and IGF-1 | Baseline Menstrual Cycle (MC) (28 days (d) or the length of 1 MC, intervention 1 (28 d or 1 MC), intervention 2 (28 d or 1 MC), intervention 3 (28 d or 1 MC), intervention 4 (28 d or 1 MC), and Post Study (days 1-7 last MC)
  Change in urine estrone-1-glucuronide (E1G ng/mL) and serum IGF-1 (ng/mL)

SECONDARY OUTCOMES:
Change in body composition | Baseline Menstrual Cycle (MC) (28 days (d) or the length of 1 MC, intervention 1 (28 d or 1 MC), intervention 2 (28 d or 1 MC), intervention 3 (28 d or 1 MC), intervention 4 (28 d or 1 MC), and Post Study (days 1-7 last MC)
  Change in percent body fat (%)
Change in body composition | Baseline Menstrual Cycle (MC) (28 days (d) or the length of 1 MC, intervention 1 (28 d or 1 MC), intervention 2 (28 d or 1 MC), intervention 3 (28 d or 1 MC), intervention 4 (28 d or 1 MC), and Post Study (days 1-7 last MC)
  fat mass (kg) and fat free mass (kg)
Change in reproductive hormones | Baseline Menstrual Cycle (MC) (28 days (d) or the length of 1 MC, intervention 1 (28 d or 1 MC), intervention 2 (28 d or 1 MC), intervention 3 (28 d or 1 MC), intervention 4 (28 d or 1 MC), and Post Study (days 1-7 last MC)
  Change in reproductive hormones sex hormone binding globulin (SHBG nmol/L)
Change in reproductive hormones | Baseline Menstrual Cycle (MC) (28 days (d) or the length of 1 MC, intervention 1 (28 d or 1 MC), intervention 2 (28 d or 1 MC), intervention 3 (28 d or 1 MC), intervention 4 (28 d or 1 MC), and Post Study (days 1-7 last MC)
  Change in reproductive hormones pregnanediol glucuronide (PdG ng/mL)
Change in metabolic hormones | Baseline Menstrual Cycle (MC) (28 days (d) or the length of 1 MC, intervention 1 (28 d or 1 MC), intervention 2 (28 d or 1 MC), intervention 3 (28 d or 1 MC), intervention 4 (28 d or 1 MC), and Post Study (days 1-7 last MC)
  Change in metabolic hormones leptin (ng/mL) and insulin-like growth factor binding protein 3 (ng/mL)
Change in metabolic hormones | Baseline Menstrual Cycle (MC) (28 days (d) or the length of 1 MC, intervention 1 (28 d or 1 MC), intervention 2 (28 d or 1 MC), intervention 3 (28 d or 1 MC), intervention 4 (28 d or 1 MC), and Post Study (days 1-7 last MC)
  Change in metabolic hormone insulin (μIU/mL)
Change in metabolic hormones | Baseline Menstrual Cycle (MC) (28 days (d) or the length of 1 MC, intervention 1 (28 d or 1 MC), intervention 2 (28 d or 1 MC), intervention 3 (28 d or 1 MC), intervention 4 (28 d or 1 MC), and Post Study (days 1-7 last MC)
  Change in metabolic hormone sex hormone binding globulin (nmol/L)
Change in metabolic hormones | Baseline Menstrual Cycle (MC) (28 days (d) or the length of 1 MC, intervention 1 (28 d or 1 MC), intervention 2 (28 d or 1 MC), intervention 3 (28 d or 1 MC), intervention 4 (28 d or 1 MC), and Post Study (days 1-7 last MC)
  Change in metabolic hormone total triiodothyronine (ng/dL)
Change in menstrual cycle phase length | Baseline Menstrual Cycle (MC) (28 days (d) or the length of 1 MC, intervention 1 (28 d or 1 MC), intervention 2 (28 d or 1 MC), intervention 3 (28 d or 1 MC), intervention 4 (28 d or 1 MC)
  Change in follicular phase length (days) and luteal phase length (days)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Williams, ScD, Principal Investigator — Penn State University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Williams NI, Reed JL, Leidy HJ, Legro RS, De Souza MJ. Estrogen and progesterone exposure is reduced in response to energy deficiency in women aged 25-40 years. Hum Reprod. 2010 Sep;25(9):2328-39. doi: 10.1093/humrep/deq172. Epub 2010 Jul 6. PMID 20605898